CLINICAL TRIAL: NCT02654210
Title: LoewenKIDS - Infections and the Development of the Immune System
Acronym: LoewenKIDS
Status: Active, not recruiting | Type: Observational
Sponsor: Helmholtz Centre for Infection Research (Other)
Collaborators: Martin-Luther-Universität Halle-Wittenberg (Other); Hannover Medical School (Other); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: HelmholtzCIfectionsRes
Record Dates: First submitted 2016-01-11; First posted 2016-01-13 (Estimated); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Infectious Diseases
Keywords: birth cohort; infectious diseases; microbiome; immune system; immune response
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasal swabs nasal: Microbiome Nasal swabs: Virus detection Stool sample: Microbiome Stool sample. Pathogen Detection Blood sample Buccal swab
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
The purpose of this study is to determine in what way infections, microbiome, and vaccinations during childhood interact in shaping the development of immunity and tolerance. The investigators collect and use data from a birth cohort focusing on infectious diseases during childhood and apply a life course perspective.

DETAILED DESCRIPTION:
The goal of the study is to capture the complete history of exposure towards microbial challenges in the first six years of life and to study interactions between different components of microbial exposure as well as effects on the development of immunity. The investigators apply a diary in which parents document symptoms of respiratory and gastrointestinal infections of their child, and collect nasal swabs and stool samples obtained on first day of symptoms. In addition, the investigators collect nasal swabs and stool samples once per year during an asymptomatic period. The investigators intend to collect venous blood from children participating in the study at the age of six years. In a subsample (called intensive subcohort), the investigators collect asymptomatic probes three monthly during the first two years of life and obtain venous blood of the children at the age of one and two years.

The study sample is 782 participants, with 285 participants in the intensive subcohort.

Symptomatic samples will be analyzed by means of multiplex polymerase chain reaction (PCR). In addition, the investigators will assess microbial compositions based on next generation sequencing and apply multiplex panels to study parameters of unspecific humoral immune response. The study will allow to assess homologous and heterologous effects of infections and vaccinations measuring specific humoral immune response. In collaboration with immunologists, immune phenotypes will be studied and functional tests will be conducted.

The investigators will use allergic dermatitis at the age of two as a primary proxy outcome and target asthma at the age of six years as a definitive clinical endpoint.

ELIGIBILITY:
Inclusion Criteria:

* newborn in a study region

Exclusion Criteria:

* parents < 18 years old
* insufficient knowledge of the German language (parents)

Ages: 1 Day to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Healthy Newborns in the Studyregions: Braunschweig, Hannover, Bremen, München, Halle (Saale), Germany
Sampling Method: Non-Probability Sample
Enrollment: 782 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2033-02 (Estimated); Study Completion 2033-02 (Estimated)

PRIMARY OUTCOMES:
Development of immune system | 15 years
  Assessment of interactions between infections, microbial colonization, vaccinations and immune response in the framework of life-course epidemiology

SECONDARY OUTCOMES:
Allergic dermatitis (yes/no) | at age of two years
  Mechanisms of microbial challenge underlying the development of atopic dermatitis in the framework of life-course epidemiology
Asthma | at age of six years
  Mechanisms of microbial challenge underlying the development of asthma in the framework of life-course epidemiology

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Mikolajczyk, Prof. Dr., Principal Investigator — Martin-Luther-University Halle-Wittenberg; Institute of Medical Epidemiology, Biometry and Informatics
Locations (2):
- Germany (2):
  - Helmholtz Centre for Infection Research, Braunschweig, Lower Saxony
  - Martin-Luther-University Halle-Wittenberg, Halle, Saxony-Anhalt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zoch B, Karch A, Dreesman J, Monazahian M, Baillot A, Mikolajczyk RT. Feasibility of a birth cohort study dedicated to assessing acute infections using symptom diaries and parental collection of biomaterials. BMC Infect Dis. 2015 Oct 22;15:436. doi: 10.1186/s12879-015-1189-0. PMID 26493700
- [Background] Gottschick C, Raupach-Rosin H, Langer S, Hassan L, Horn J, Dorendorf E, Caputo M, Bittner M, Beier L, Rubsamen N, Schlinkmann K, Zoch B, Guzman CA, Hansen G, Heselich V, Holzapfel E, Hubner J, Pietschmann T, Pieper DH, Pletz M, Riese P, Schmidt-Pokrzywniak A, Hartwig S, von Kaisenberg C, Aydogdu M, Buhles M, Dressler F, Eberl W, Haase R, Edler von Koch F, Feidicker S, Frambach T, Franz HGB, Guthmann F, Koch HG, Seeger S, Oberhoff C, Pauker W, Petry KU, Schild RL, Tchirikov M, Rohrig E, Karch A, Mikolajczyk R. Cohort Profile: The LoewenKIDS Study - life-course perspective on infections, the microbiome and the development of the immune system in early childhood. Int J Epidemiol. 2019 Aug 1;48(4):1042-1043h. doi: 10.1093/ije/dyz001. No abstract available. PMID 30815674
- [Background] Langer S, Horn J, Gottschick C, Klee B, Purschke O, Caputo M, Dorendorf E, Meyer-Schlinkmann KM, Raupach-Rosin H, Karch A, Rubsamen N, Aydogdu M, Buhles M, Dressler F, Eberl W, Koch FEV, Frambach T, Franz H, Guthmann F, Guzman CA, Haase R, Hansen G, Heselich V, Hubner J, Koch HG, Oberhoff C, Riese P, Schild R, Seeger S, Tchirikov M, Trittel S, von Kaisenberg C, Mikolajczyk R. Symptom Burden and Factors Associated with Acute Respiratory Infections in the First Two Years of Life-Results from the LoewenKIDS Cohort. Microorganisms. 2022 Jan 5;10(1):111. doi: 10.3390/microorganisms10010111. PMID 35056559
- [Derived] Lincetto C, Romero-Saavedra F, Laverde D, Lincetto R, Meyer-Buehn M, Klee B, Gottschick C, Mikolajczyk R, Huebner J, Schober T. Detection of enteric pathogens in young children before and during acute gastroenteritis: results from a prospective German birth cohort study (LoewenKIDS). Infection. 2025 Oct 20. doi: 10.1007/s15010-025-02670-1. Online ahead of print. PMID 41114888
- See also: Study website [click here to get more information (German only)] — http://www.loewenkids-study.de